CLINICAL TRIAL: NCT04874051
Title: Sensor-Based Analysis And rehabiLitation of bAlance in Neurological Diseases: a multiCentric randomizEd Clinical Trial
Brief Title: Sensor-based Assessment and Rehabilitation of Balance in Neurological Diseases
Acronym: BALANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: IRCCS San Raffaele (Other); Istituti Clinici Scientifici Maugeri SpA (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1099/IRCCS San Camillo
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Multiple Sclerosis; Parkinson Disease
Keywords: Balance; Sensor-based rehabilitation; Virtual Reality
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The experimental group is treated through a sensor-based devices in a virtual environment, while the control group is treated through conventional physiotherapy for balance rehabilitation
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): In the EG the subjects will perform balance exercises using the OAK system under the supervision of a trained physiotherapist. The treatment will last 3 weeks with daily sessions of 60 minutes, 5 times per week.
  Interventions: Device: Experimental Group
- Control Group (CG) (Active Comparator): In the CG the subjects will be asked to perform conventional balance exercises under the supervision of a physiotherapist. The treatment will last 3 weeks with daily sessions of 60 minutes, 5 times per week.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Experimental Group — The experimental treatment will be provided by means of the OAK system. This device consists of 1 cabinet with 2 independent balance boards, 2 monitors (one for the physiotherapist and one for the patient) and 3 wireless IMUs (one for the left lower limb, one for the right lower limb and one for the trunk). The 2 balance boards provide body weight transfer exercises, while the wireless motion sensors provide one leg stance exercises or trunk exercises in a virtual environment.
  Arms: Experimental Group (EG)
Other: Control Group — The Control Group will perform conventional balance exercises similar to the exercises provided with the OAK system.
  Arms: Control Group (CG)

SUMMARY:
Balance impairment is one of the most common disorders due to a neurological diseases. Sensor-based technologies may be useful for falls prevention and balance recovery during patients hospitalization. OAK Elderly Care System (Khymeia Group, Noventa Padovana, Italy) allows the assessment of fall risk, the centre of pressure and the execution of balance exercises in a virtual environment.

DETAILED DESCRIPTION:
The aim of the study is to compare the therapy provided by means of the OAK Elderly Care System with conventional physiotherapy for balance rehabilitation in patients affected by stroke, Multiple Sclerosis (MS) and Parkinson Disease (PD).

OAK Elderly Care System consists of two independent balance boards and three sensors for the kinematic tracking of the trunk and lower limbs. These components allow the assessment of the centre of pressure and the execution of exercises in a virtual environment.

120 patients (40 stroke, 40 MS, 40 PK) hospitalized at 4 different italian hospitals, were enrolled according to inclusion and exclusion criteria and randomly assigned to two groups (i.e. intervention group, control group). Intervention group received 1 daily hour of technology-based treatment, while the control group underwent 1 daily hour of physiotherapy for balance rehabilitation, in addiction to 1 hour of conventional physiotherapy. Both treatments lasted 15 sessions. Before and after treatment balance, walking, daily living autonomy and pathology-specific features were assessed.

ELIGIBILITY:
Inclusion Criteria:

Common criteria:

* Berg Balance Scale < 50/56;
* Ability to maintain the standing position with o without one support for 1 minute;
* Functional Independence measure < 100/126;
* Barthel Index < 80/100.

Stroke:

* Single ischemic stroke;
* Lesion occured after 2 and within 18 months;
* National Institute of Health Stroke Scale ≤ 14.

Parkinson:

* 1.5 < Hoehn & Yahr < 3;
* Subitem "freezing when walking"of the UPDRS ≤ 2.

Multiple Sclerosis:

* Relapsing remitting or secondary progressive Multiple Sclerosis;
* Expanded Disability Status Scale ≤ 6.5.

Exclusion Criteria:

* Untreated epilepsy;
* Major depressive disorder;
* Fractures;
* Dementia;
* Ideomotor Apraxia;
* Neglect;
* Severe impairment of verbal comprehension;
* Severe acoustic and visual disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Change from baseline Berg Balance Scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means better outcome (minimum score = 0, maximum score = 56).

SECONDARY OUTCOMES:
Number of falls during the last year | Change from baseline number of falls during the last year scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions).
Functional Ambulation Classification (FAC) | Change from baseline Functional Ambulation Classification at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means better outcome (minimum score = 0, maximum score = 5).
Activities specific-Balance Confidence scale (ABC) | Change from baseline Activities specific-Balance Confidence scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means better outcome (minimum score = 0, maximum score = 100).
Functional Independence Measure (FIM) | Change from baseline Functional Independence Measure at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means better outcome (minimum score = 0, maximum score = 126).
Barthel Index (BI) | Change from baseline Barthel Index at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means better outcome (minimum score = 0, maximum score = 100).
National Institution of Health Stroke Scale (NIHSS) | Change from baseline National Institute of Health Stroke Scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means worse outcome (minimum score = 0, maximum score = 42).
Unified Parkinson's Disease Rating Scale (UPDRS) | Change from baseline Unified Parkinson's Disease Rating Scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means worse outcome (minimum score = 0, maximum score = 147).
Hoehn & Yahr Scale (H&Y) | Change from baseline Hoehn & Yahr Scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means worse outcome (minimum score = 0, maximum score = 5).
Kurtzke Extended Disability Status Scale (EDSS) | Change from baseline Kurtzke Extended Disability Status Scale at the end of the therapy (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). A higher score means worse outcome (minimum score = 0, maximum score = 10).

OTHER OUTCOMES:
Instrumental assessment | Change from baseline BBS at the end of the therapy (three weeks thereafter)
  The OAK system will record the changes of the center of pressure during 30 seconds, with relaxed arms and eyes open.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, PhD, Principal Investigator — San Camillo IRCCS
Locations (5):
- Italy (5):
  - IRCCS Fondazione Mondino, Pavia
  - IRCCS ICS Maugeri Spa SB, Pavia
  - IRCCS San Raffaele Pisana, Rome
  - IRCCS Fondazione Santa Lucia, Rome
  - San Camillo IRCCS, Venice